CLINICAL TRIAL: NCT02917603
Title: Shared Decision Making to Improve Palliative Care in the Nursing Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Debra Parker Oliver, Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2003012
Record Dates: First submitted 2016-09-23; First posted 2016-09-28 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): These family members and residents will use web conferencing technology to attend their quarterly care conferences
  Interventions: Behavioral: Web Conferencing
- Control (No Intervention): These family and residents will receive usual care

INTERVENTIONS:
Behavioral: Web Conferencing — Individuals will communicate with the nursing home team via web conferencing during quarterly care conference
  Arms: Intervention

SUMMARY:
Twenty-eight percent of Americans over the age of 65 die in a nursing home. Research has found the quality of care of end-of-life care in nursing homes to have many challenges. It has also been documented that family members, especially those living at a distance, want to be involved in the care of their resident and family support can be beneficial to residents. Family members' involvement in decision-making in the nursing home setting improves outcomes for residents with life-limiting illnesses. Shared decision-making (SDM) is a process wherein a healthcare choice is jointly made by a healthcare provider and a resident or resident's proxy, often a family member. This proposal seeks to facilitate SDM among family members, residents with life-limiting illnesses (who are not enrolled in hospice), and the nursing home care team. The overall research question (RQ) asks: To what extent are outcomes for family member and residents with life limiting illnesses associated with SDM via web-conferencing in the nursing home? The overall hypothesis (H) is that SDM among family members, residents (when possible), and skilled nursing home staff via web-conferencing will improve outcomes for family members and residents with life-limiting illnesses. This is an exploratory mixed methods randomized clinical trial pilot to test the effect of shared decision making using web-based conferencing on the depression and burden of family members and the pain of nursing home residents.

DETAILED DESCRIPTION:
Twenty-eight percent of Americans over the age of 65 die in a nursing home. Research has found that the quality of care at the end of life in these facilities is less than adequate. While some residents improve their care with the use of the Hospice Medicare benefit, considerable barriers remain for the majority of nursing home residents who do not enroll in hospice but have a serious illness. This project focuses on improving palliative care for geriatric nursing home residents who are not receiving hospice care. Two systematic reviews of end-of-life care in nursing homes found challenges in symptom burden, including unmanaged pain, inadequate discussions regarding goals of care and advance directives, poor communication, unmet family expectations, and inadequate staff education.

Residents' values, beliefs, and goals are often unknown by nursing home staff. Dementia, illness, or poor communication may prevent residents from articulating their wishes regarding care. In many cases, family members can act as mediators between the resident and staff as plans of care are developed and decisions are made. Despite the desire to remain involved in care of the nursing home resident, many family members are unable to be physically present in the nursing home and experience loss of control, dis-empowerment, and guilt. As frailty increases and goals of care become increasingly palliative, the frustrations and burdens for families can worsen. Family members, especially those living at a distance, want to be involved in the care of their resident, and their involvement in decision-making can improve outcomes for residents with serious illnesses.

This project facilitates SDM (shared decision making) among family members, residents with serious illnesses (not enrolled in hospice), and the nursing home care team. Based on a family-identified need, this proposal facilitates SDM among family members, residents with serious illnesses (not enrolled in hospice), and the nursing home care team.

ELIGIBILITY:
Inclusion Criteria:

* Residents: Residents of The Bluffs nursing home, Columbia Missouri, over the age of 65, have at least one family member who agrees to participate, and have a serious life limiting illness. Residents enrolled in hospice or admitted to post hospital short term nursing home stay are excluded from participation.
* Family Members: Identified family member by a resident or nursing home staff at The Bluffs, over the age of 18, without cognitive impairment, and with access to a computer, tablet, or smartphone device.

Exclusion Criteria:

* Residents enrolled in hospice can not participate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Oliver, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- The Bluffs, Columbia, Missouri, United States

REFERENCES:
- [Derived] Oliver DP, Rolbiecki AJ, Washington K, Kruse RL, Popejoy L, Smith JB, Demiris G. A Pilot Study of An Intervention to Increase Family Member Involvement in Nursing Home Care Plan Meetings. J Appl Gerontol. 2021 Sep;40(9):1080-1086. doi: 10.1177/0733464820946927. Epub 2020 Aug 13. PMID 32787506

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 20 | 20
Completed | 19 | 16
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Customized [Mean (Standard Deviation); unit: Years]
  Mean Age at consent | 55.7 (8.4) | 57.2 (9.5) | 56.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 20 | 19 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Anxiety (GAD-7) [Mean (Standard Deviation); unit: Score on a scale] — Participants complete and each question is rated 0 (not at all)- 3 (nearly every day) for total scores of 0-21. 5,10,15 indicate mild, moderate, or severe anxiety. A score of 10 or higher indicates clinically significant anxiety.
  Score on a scale | 2.10 (3.34) | 2.10 (2.86) | 2.10 (3.07)
Depression (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] | 1.50 (1.47) | 2.55 (3.63) | 2.03 (2.79)
Burden (Zarit) [Mean (Standard Deviation); unit: score on a scale] — Zarit Burden Interview is a scale. Each question is scored 0 (best) to 4 (worse). Response options for each item range from 0-4, and total scores range from 0-88, with higher scores indicating greater self-reported burden
  score on a scale | 2.45 (2.37) | 3.7 (3.6) | 3.08 (3.08)
Caregiver Quality of Life (CQLI-R) [Mean (Standard Deviation); unit: units on a scale] — The instrument rates caregiver quality of life on a scale of 0-9 with 0 being the best quality of life and 9 being the worse. It has four questions each for a total score of 0-36. The higher the score the worse the quality of life
  units on a scale | 33.75 (5.14) | 30.95 (7.04) | 32.35 (6.25)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Mean Patient Health Questionaire 9 Score From Baseline
Description: 9 questions that indicate depression- taken at 30 days-Scale is 0-27 with higher values representing more depression. Measure collected every 30 days. Analysis is a comparison of means between the last measure taken and the baseline scores- with an overall average then computed.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 20
units on a scale | .74 (1.19) | 3.38 (3.5)
Statistical Analysis 1: Comparison: Intervention vs Control; The null hypothesis is that the mean differences between baseline and last measure in the PHQ- 9 score will not differ between groups. Study is powered a two-tailed test of significance, allowing the detection of a significant difference in either direction and the following assumptions: expected difference in PHQ-9 is 5 points, the documented clinically significant effect;78 (2) the variance of scores is 5.33; (3) error protection: α =.10, β = .20 and, (4) anticipated attrition of 15%; Test type: Equivalence — Null hypothesis is that there would be no mean difference between baseline and last measure between intervention and control groups with p<.05; p < .009, t-test, 2 sided; Mean Difference (Net) = .12

2. Secondary Outcome: Zarit Burden Interview
Description: Family members will report which of their responsibilities are perceived as burdensome. Response options for each item range from 0-4, and total scores range from 0-88, with higher scores indicating greater self-reported burden. Total score computed with an average score response.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 19 | 16
units on a scale | 3.16 (2.63) | 4.25 (4.93)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Equivalence — Null hypothesis is there will be the mean differences between baseline scores will be the same between groups. Study powered after primary outcome measure; p < .21, t-test, 2 sided; Mean Difference (Net) = .46

3. Secondary Outcome: Generalized Anxiety- 7
Description: 7 questions that measure family member anxiety. It has 7 items and is scored 0-21 with a higher number representing greater anxiety. A total score is computed.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 19 | 16
score on a scale | .63 (.96) | 2.06 (2.72)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p < .06, t-test, 2 sided; Mean Difference (Net) = 1.02

4. Secondary Outcome: Caregiver Quality of Life
Description: 4 questions pertaining to family quality of life. There are 4 items each scored 0-9 with a total score of 0 to 36 and higher scores representing poorer quality of life.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 19 | 16
units on a scale | 33.79 (4.21) | 32.06 (7.89)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p < .73, t-test, 2 sided; Mean Difference (Net) = .23

ADVERSE EVENTS:
Time Frame: 1 year 7 months
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2016-12-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT02917603/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2015-11-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT02917603/Prot_SAP_001.pdf